CLINICAL TRIAL: NCT04075357
Title: Amniotic Membrane Transplantation for Carpal Tunnel Syndrome Treatment: One-year Follow-up
Brief Title: Amniotic Membrane in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2016/10/04
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Amniotic membrane transplantation
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The patients underwent conventional CTS surgery
- Experimental (Experimental): The patients underwent conventional CTS surgery and transplantation of amniotic membrane
  Interventions: Other: Amniotic membrane transplantation

INTERVENTIONS:
Other: Amniotic membrane transplantation — Amniotic membrane was located over median nerve during surgery of CTS, prior of closing.
  Arms: Experimental

SUMMARY:
Carpal Tunnel Syndrome (CTS) is the most frequent mononeuropathy. CTS is more frequent in females than in males, it has been associated to work activities, hormone exposure and obesity. Although its primary treatment is conservative, there is strong evidence that patients who retard surgery are more prone to develop worse outcomes. Surgery to treat CTS consists in liberating carpal tunnel in order to ameliorate median nerve symptoms; however, more than 20% of patients who undergo surgery have recurrent CTS (RCTS). RCTS is due to a fibrotic process in the site of the surgery. Amniotic membrane (AM) is the inner layer of the placenta which has been used to treat different pathologies. AM transplantation (AMT) has demonstrated to significantly inhibit inflammation and fibrosis. Therefore, the aim of the present study was to determine the effect of AMT in CTS surgery. The present is a randomized, open labeled, controlled clinical study. The investigators included patients with recent diagnosis of CTS and divided into two groups. The experimental group received AMT concomitantly with conventional surgery; whilst, the control group received only the conventional surgery. Clinical status of patients measured with the BCTQ questionaire was the main outcome. Both groups showed similar BCTQ punctuation at the beginning of the study. However, the results of the experimental group were significantly better than those from the control group through time, until the finish of the study. None of the patients presented complications or adverse effects related to the AMT. These results indicate that AMT is a secure and suitable treatment for CTS presenting better clinical outcomes at one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent CTS diagnosis
* Patients that undergo CTS surgery
* Patients that accept to participate in the study
* Patients that sign informed consent

Exclusion Criteria:

* Patients with recurrent CTS diagnosis;
* Patients with concomitant hand/arm comorbidities
* Patients with any systemic disease that comprises muscles and bones
* Collagenopathies
* Systemic lupus erythematosus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
BCTQ | Through study completion, an average one year
  The Boston Carpal Tunnel Questionnaire (BCTQ) is a disease-specific measure of self-reported symptom severity and functional status. It is frequently used in the reporting of outcomes from trials into interventions for carpal tunnel syndrome.
  It has two distinct scales, the Symptom Severity Scale (SSS) which has 11 questions and uses a five-point rating scale and the Functional Status Scale (FSS) containing 8 items which have to be rated for degree of difficulty on a five-point scale. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be published in a Journal. Therefore it will be supplied elsewhere.

REFERENCES:
- [Derived] Buentello-Volante B, Molina-Medinilla M, Aguayo-Flores E, Magana-Guerrero FS, Garfias Y. Comparison of amniotic membrane transplantation and carpal tunnel syndrome release surgery (CTRS) and CTRS alone: Clinical outcomes at 1-year follow-up. J Tissue Eng Regen Med. 2020 May;14(5):714-722. doi: 10.1002/term.3033. Epub 2020 Mar 24. PMID 32174033